CLINICAL TRIAL: NCT03505411
Title: The Influence of Melatonin Supplementation in the Group of Persons Performing Competitive Sport.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Jolanta Czuczejko, Assistant professor, Nicolaus Copernicus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KB 586/2009
Record Dates: First submitted 2018-03-28; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Antioxidants; Oxidative Stress; Inflammation; Lipid Peroxidation
Keywords: Melatonin; Glutathione; Glutathione peroxidase; Malondialdehyde; Isoprostanes; anti-ox-LDL; Superoxide dismutase; Glutathione reductase; Interleukin-6; C-reactive protein; Autonomic nervous system
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- melatonin, submaximal effort (Experimental): 1 arm 5 mg melatonin 1 hr before bedtime for 30 days
  Interventions: Dietary Supplement: melatonin supplementation

INTERVENTIONS:
Dietary Supplement: melatonin supplementation

SUMMARY:
The research aims to determine the impact of 30-day supplementation of melatonin on the antioxidative defense mechanisms and the release of markers of oxidative stress and inflammation in rowers and footballers undergoing training of submaximal intensity.

DETAILED DESCRIPTION:
Athlete's body, by its high oxygen demand and increased aerobic metabolism, is exposed to the formation and oxidizing action of reactive oxygen species (ROS). Imbalance between the mechanisms of ROS generation and antioxidative defense of the body can lead to oxidative stress expressed by elevated concentrations of lipid peroxidation products, such as malondialdehyde, isoprostanes (8-iso-PGF2α), oxidized low-density lipoprotein molecules (ox-LDL). The body's defense against ROS includes two systems: nonenzymatic and enzymatic. Small-molecule antioxidants include reduced glutathione (GSH). Due to the presence of -SH groups, glutathione has strong reductive properties. The compound is a substrate for glutathione peroxidase (GSH-Px) which decomposes hydrogen peroxide and organic peroxides. Among antioxidant enzymes are also: superoxide dismutase (Cu-Zn-SOD, scavenges superoxide anion radical), catalase (CAT, reduces hydrogen peroxide), and glutathione reductase (GR, reduces oxidized glutathione). Another well-known small-molecule antioxidant is melatonin, hormone of the pineal gland. It has been demonstrated that this compound can reduce hydrogen peroxide, scavenge hydroxyl radical and deactivate nitric oxide radical.

Another manifestation of disruption of homeostasis in the body of a professional athlete are enhanced inflammatory processes. This can be explained by the fact that during physical effort of varied intensity, increased activity of myeloperoxidase and higher levels of mRNA for tumor necrosis factor, interleukin-1 and -6 are observed. Interleukin-6, also known as myokine, is a particularly important marker of intense physical effort released from damaged muscles. Myokine is also the main upregulator of the synthesis of C-reactive protein (CRP) in the liver, hence measuring the concentration of the protein can indicate the intensity of inflammatory processes in an athlete's body. It has been demonstrated that melatonin, in addition to its hormonal and antioxidant properties, can modulate inflammatory processes by reducing the synthesis of proinflammatory cytokines.

Taking into account the multidirectional function of melatonin, it seems interesting to establish the impact of 30-day supplementation of this hormone on the antioxidative defense mechanisms and the release of markers of oxidative stress and inflammation in rowers and footballers undergoing training of submaximal intensity.

ELIGIBILITY:
Inclusion Criteria:

* sign informed consent form for participation in the study

Exclusion Criteria:

* diseases
* the participants will not be minor and incapacitated persons, soldiers, prisoners and persons dependent in any way from the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-01-15 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of oxidative stress parameters and inflammatory markers concentration before melatonin administration, at baseline. | 1 day
  The study was conducted in football players and rowers and the control group. Samples of blood from the basilic vein were taken once, from both the control group and the athletes at baseline. In blood serum, the ELISA method was used to determine the concentrations of melatonin, isoprostanes (8-iso-PGF2α), anti-ox-LDL antibodies, interleukin-6 and C-reactive protein (CRP). In red blood cells, the concentration of reduced glutathione (GSH), thiobarbituric acid reactive substances (malondialdehyde, MDA) were determined and the activity of glutathione peroxidase (GSH-Px), cytoplasmic superoxide dismutase (SOD-1) and glutathione reductase (GR) were determined.

SECONDARY OUTCOMES:
Changes in oxidative stress parameters and inflammatory markers concentration afer 30 days of melatonin administration in athletes. | 30 day
  After 30 days of melatonin supplementation, samples of blood from the basilic vein were taken only from athletes, once, in the same day. In biochemistry laboratory, in blood serum, the ELISA method was used to determine the concentrations of melatonin, isoprostanes (8-iso-PGF2α), anti-ox-LDL antibodies, interleukin-6 and C-reactive protein (CRP). In red blood cells, the concentration of reduced glutathione (GSH), thiobarbituric acid reactive substances (malondialdehyde, MDA) were determined and the activity of glutathione peroxidase (GSH-Px), cytoplasmic superoxide dismutase (SOD-1) and glutathione reductase (GR) were determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Czuczejko, Principal Investigator — Department of Positron Emission Tomography and Molcecular Diagnostics, Collegium Medicum of Nicolaus Copernicus University

IPD SHARING:
Plan to Share IPD: No
There is no the IPD sharing plan.